CLINICAL TRIAL: NCT06266078
Title: A Human Factors Simulation Study Protocol for the Assessment of Usability of Innovative Personal Protective Equipment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Caroline Lopes Ciofi Silva, Professor, University of Campinas, Brazil
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Device Feasibility
Other Study IDs: School of Nursing
Record Dates: First submitted 2024-02-02; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Personal Protective Equipment
Keywords: Ergonomics; Personal Protective Equipment; Simulation-Based Research
MeSH Terms: interventions — N95 Respirators

STUDY DESIGN:
Intervention Model Description: Firstly, a minimum of 14 experts will validate the content, using the Delphi technique of two tools (A) The innovative PPE assessment tool; and B) the simulation scenario script.
  After reaching consensus among the experts, the protocol will be piloted. Two identical sessions will be conducted using the cross-over method with all participants, so that the same participant performs the tasks using the innovative PPE and the comparative PPE, allowing the participants compare characteristics of both PPE. The PPE use sequence and the PPE type will be randomized to minimize biases. Between both sessions there will a 30-minute break for the participants.
  For the purpose of the development and piloting of this simulation protocol, the innovative PPE were selected according to compliance with the specifications required by the World Health Organization. It will enrolled 36 healthcare workers in piloting test.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Innovative PPE (Experimental): The healthcare workers will perform tasks using non-traditional personal protective equipments.
  Interventions: Device: Innovative PPE
- Traditional PPE (Active Comparator): The healthcare workers will perform tasks using traditional personal protective equipments.
  Interventions: Device: Traditional PPE

INTERVENTIONS:
Device: Innovative PPE — The healthcare workers will perform tasks using innovative personal protective equipments, such as LightWeight Powered Air-Purifying Respirator (PAPR) or other type of PAPR and a Sealed coverall
  Other Names: PAPR and Coverall
  Arms: Innovative PPE
Device: Traditional PPE — The healthcare workers will perform tasks using usual personal protective equipments, such as N95 mask plus Faceshield and waterproof apron.
  Other Names: N95 Mask + Faceshield and Apron
  Arms: Traditional PPE

SUMMARY:
Background: Many factors influence Personal Protective Equipment (PPE) compliance for use in health care, specifically the PPE usability and related human factors. It is known that issues related to the usability of new technologies, including professional behavioral and attitudinal patterns, the technologies adoption within the workflow and teamwork strengths can be investigated by using Simulation-Based Research (SBR) before its implemented. This study aims to develop and validate a simulation protocol for the assessment of human factors and usability of innovative PPEs used in critical care units. The ultimate goals is to define a standard method for PPEs assessment and comparison worldwide. Method: methodological study with a quantitative approach to be carried out in two phases: a) development and validation by experts of a simulation protocol; b) piloting of the simulation protocol. For the protocol validation phase, 14 experts with experience in the themes of infection prevention and control or clinical simulation will be included. The experts will be invited via email and will assess the simulation protocol content using the criteria of pertinence, clarity and relevance. To ensure that the simulation protocol is feasible and reliable, a piloting phase will take place at the simulation center in São Paulo and 36 health professionals with work experience in critical care units will be included. The health professionals will perform specific tasks assigned to them, wearing pre-defined PPEs in each simulation round. Errors and difficulties during PPE assembly, donning and doffing; performance of individual and team activities, as well as communication problems and self-contamination risk, will be observed during the tasks. At the end of the simulation round, the participants will take part in a debriefing, where they will answer questionnaires about comfort, perception of safety, thermal sensations, usability and perceived workload related to the PPE used. Content validity index (CVI) and intraclass correlation coefficient (ICC) will be calculated. This study protocol was approved by the Research Ethics Committee of the School of Nursing, University of São Paulo. The informed consent form will be applied both to the experts and to the health care workers.

DETAILED DESCRIPTION:
The study design is a methodological study with a quantitative approach, consisting of two phases. In phase 1 we will perform a virtual development and content validation by experts, of an innovative PPE assessment simulation. In phase 2 we will pilot the simulation protocol. Phase 2 will be conducted in the simulation center of the School of Nursing, University of São Paulo.

Phase 1 - For content validation, a minimum of 14 experts will be included [21]. The experts shall have experience in the themes of infection prevention and control (IPC) and simulation studies to validate the data collection tool. Considering that the intention is for the simulation protocol to be applicable in different countries, experts working in Brazil and in foreign countries will be included. The experts must be fluent in the Portuguese or English languages, have a minimum degree of specialization in the health areas, and have academic experience, as evidenced by publications in indexed scientific journals over the last three years. The search for experts working in Brazil will be performed through a platform of the researchers' resumes, available on the National Council for Scientific and Technological Development (CNPq) portal, as well as in reference lists of scientific papers on the theme. Experts working in other countries will also be selected through the reference list of scientific papers and after analyzing the information recorded in the Open Researcher and Contributor platform: ID (ORCID).

Phase 2 - The simulation protocol piloting will include HCW with work experience in critical care (intensive care units and emergency department) for adult patients, from the following professional categories: physicians, nurses, nursing technicians and physiotherapists, with at least one year of experience, and regardless of gender. Professionals taking part in simulation studies in the last year, with similar content, will be excluded. The convenience sample will be invited by word of mouth and by means of posters in selected hospitals in São Paulo.

After reaching consensus regarding the clinical simulation script among the experts, the protocol will be piloted. After accepting to take part in the research by signing a written consent form, the participants will be emailed informational materials about the activities that will be performed and instructional material about the PPE items that will be used.

Two identical sessions will be conducted using the cross-over method with all participants, so that the same participant performs the tasks using the innovative PPE and the comparative PPE, allowing the participants compare characteristics of both PPE. The PPE use sequence and the PPE type will be randomized to minimize biases. Between both sessions there will a 30-minute break for the participants.

ELIGIBILITY:
Phase 1 - For content validation, a minimum of 14 experts will be included.

Inclusion criteria:

* Have experience in the themes of infection prevention and control (IPC) and simulation studies;
* Work in Brazil and in foreign countries;
* Be fluent in the Portuguese or English languages;
* Have a minimum degree of specialization in the health areas;
* Have academic experience, as evidenced by publications in indexed scientific journals over the last three years.

Exclusion criteria - None

Phase 2 - For simulation protocol piloting, NINE participants from each professional category will be included

Inclusion Criteria

* Healthcare workers with experience in critical care (intensive care units and emergency department) for adult patients;
* Working as physicians, nurses, nursing technicians and physiotherapists, regardless of gender;
* With at least one year of experience.

Exclusion Criteria:

- Healthcare workers taking part in simulation studies in the last year, with similar content.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Content Validity of the items included in the "Innovative PPE assessment tool" and in the "Simulation scenario script" | During validation phase, the experts will record their answers by email. Up to three consultation rounds will be conducted.
  The experts will assess the documents sent by email and will be instructed to record their opinions, answering in a five-point Likert-type scale ("Strongly agree", "Partially agree", "Neither agree nor disagree", "Partially disagree" and "Strongly disagree") whether they agree or disagree regarding the pertinence, clarity and relevance of each item. The experts' responses will be analyzed and the Content Validity Index (CVI) as well as the Intraclass Correlation Coefficient (ICC) will be calculated.
Errors during PPE assembly/preparation, donning and doffing | Once for each PPE, while the participant is performing the task in the simulation session
  The researcher will observe the participants performing the clinical tasks and will record the following data:
  * Were there any errors while assembling/preparing the PPE? Yes or No
  * Did the participant need help while assembling/preparing the PPE? Yes or No
  * Were there any errors while donning? Yes or No
  * Did the participant need help while donning? Yes or No
  * Were there any errors while doffing? Yes or No
  * Did the participant need help while doffing? Yes or No
Communication impairments while using PPE | Once for each PPE, while the participant is performing the task in the simulation session
  The researcher will observe the participants performing the clinical tasks and will record the following data:
  * Were there any problems with verbal communication related to PPE use? Yes or No
  * Did the participants have PPE-related hearing difficulties while performing the tasks? Yes or No
Self-contamination risk in the professional while using and doffing the PPE | Once for each PPE, after removing it
  A fluorescent tracer will be used, which is a transparent dye that only becomes visible when exposed to ultraviolet light. The solution is an abrasion-resistant solution but can be easily removed with a standard cleaning procedure. The tracer will be applied to the PPE used before the start of simulation activities. After the PPE doffing, the researchers will directly visualize the body areas contaminated with the dye, in a dark room, using ultraviolet light and will note this in the data collection tool. The number of contaminated body areas will be considered.
  The researcher will observe the body areas and will record the following data:
  - Did the participant have any of body area contaminated with the dye after doffing? Yes or Not. If yes, register which areas have been contaminated.
Influence of PPE on individual performance | Once for each PPE, while the participant is performing the task in the simulation session
  The researcher will observe the participants performing the clinical tasks and will record the following data:
  * Were there any errors related to PPE while performing the tasks? Yes or No
  * Did the participant need PPE-related help while performing the tasks? Yes or No
Influence of PPE on team performance and behavioral changes | Once for each PPE, while the participants are performing the task in the simulation session
  The researcher will observe the participants performing the clinical tasks and will record the following data:
  * Were there any problems related to the assistance provided by the team to the simulated patient? Yes or No
  * Were there any difficulties related to team performance to meet the objectives proposed? Yes or No
Changes in mobility and comfort while using PPE | Once, during the debriefing period, after the participants performing the tasks
  The participants will answer the following questions, by filling in a specific form, after finishing the clinical tasks:
  * Did you notice any innovative PPE-related movement restriction while performing your tasks in the simulation setting? ( ) Frequently; ( ) Sometimes; ( ) No
  * In relation to comfort and compared to traditional PPE, the innovating PPE is: ( ) More comfortable; ( ) As comfortable as traditional; PPE ( ) Less comfortable
Thermal sensations | Once, during the debriefing period, after the participants performing the tasks
  The participants will answer the following question, by filling in a specific form, after finishing the tasks:
  - Did you feel heat or other kind of thermal discomfort while performing your tasks using the innovative PPE? ( ) Frequently; ( ) Sometimes; ( ) No
Perception regarding safety and satisfaction of the PPE user | Once, during the debriefing period, after the participants performing the tasks
  The participants will answer the following question, by filling in a specific form, after finishing the clinical tasks:
  * In relation to the safety perception, did you feel completely safe when using the innovative PPE? ( ) Agree; ( ) Indifferent; ( ) Disagree
  * What was your degree of satisfaction when using the innovative PPE? ( ) Satisfied; ( ) Indifferent; ( ) Unsatisfied
Perceived workload | Once, during the debriefing period, after the participants performing the tasks
  It will be used the "NASA Task Load Index" which is an instrument that was developed by Hart and Staveland (1988) and recently translated and validated from English into Brazilian Portuguese. Three of the six dimensions refer to aspects or requirements imposed by the subject (mental, physical and temporal demand) and the other three to the subject-task interaction (performance, effort and frustration).
Usability | Once, during the debriefing period, after the participants performing the tasks
  It will be used the System Usability Scale (SUS) which is a five-point Likert-type scale consisting of 10 assertions and which provides an overview of the user's subjective evaluations about usability of a given system, technology or product. For the current study, the instrument used will be a version of the scale translated and validated for Portuguese

SECONDARY OUTCOMES:
Complementary Content Analysis - qualitative data | Two focus group meetings will be held, one with the Brazilian experts and another with the international experts, up to a month after the end of the pilot test.
  Once the simulation protocol piloting phase is finished, the images obtained will be edited and will be sent to the same experts who took part in the first evaluation (Validation phase) of the simulation script for them to record their opinions on the piloting.
  After the experts analyze the images, two focus group meetings will be held, one with the national experts and another with their international counterparts, through an online meeting to discuss and reach agreements about the data collection script and the simulation protocol script. The following question will guide the focus group discussion: "In the format in which they were prepared, does the data collection script and the simulation protocol allow adequately assess innovation in PPE?".
  The comments from experts during the focus group will be analyzed considering following the technique proposed by Bardin (2011), in view of the Consolidated Framework for Implementation Research (CFIR) constructs.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Clara Padoveze, PhD, Study Chair — University of Sao Paulo

IPD SHARING:
Plan to Share IPD: No
Identified or identifiable data and/or information will not be provided to people who are not part of the research team. For greater data security, the following measures will be adopted: participants will be identified with letters and the database will be password-protected, with access restricted to members of the research team.